CLINICAL TRIAL: NCT04011878
Title: Histopathological Examination of Iris Tissue in Buphthalmos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Prof., Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2323299
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Iris Disease
MeSH Terms: conditions — Iris Diseases | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- isolated trabeculodysgensis (Experimental): etiology of primary congenital glaucoma
  Interventions: Procedure: Combined trabeculotomy trabeculectomy with mitomycin C

INTERVENTIONS:
Procedure: Combined trabeculotomy trabeculectomy with mitomycin C — Combined trabeculotomy trabeculectomy with mitomycin C with histopathological examination of the peripheral iris tissue specimen of all cases

SUMMARY:
To revise the etiology of the primary congenital glaucoma in some infants.

DETAILED DESCRIPTION:
Combined trabeculotomy trabeculectomy with mitomycin C was done in 11 eyes. Histopathological examination of the peripheral iris tissue specimen was done in all cases.

ELIGIBILITY:
Inclusion Criteria:

* infants under age of 2 years
* 1ery glaucoma

Exclusion Criteria:

* infants more than 2 years
* 2ery glaucoma
* previous glaucoma surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
fibrovascular membrane over iris surface | 6 month
  angle closure by a fibrovascular tissue proliferation over the trabecular meshwork in the anterior chamber angle.

IPD SHARING:
Plan to Share IPD: No